CLINICAL TRIAL: NCT04235803
Title: Telemedicine Follow-up for Routine, Low-Risk Oculoplastic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Eye plastic telemedicine
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Eyelid Diseases; Ptosis, Eyelid; Blepharoptosis; Dermatochalasis; Ectropion; Entropion; Eyelid Tumor; Skin Cancer, Eyelid; Floppy Eyelid Syndrome
Keywords: Oculoplastic; Eye plastic; Eyelid surgery; Telemedicine; Remote follow-up; Remote visit; Blepharoplasty; Ptosis repair; External levator resection; Internal levator resection; Ectropion repair; Entropion repair
MeSH Terms: conditions — Eyelid Diseases; Blepharoptosis; Cutis Laxa; Ectropion; Entropion; Eyelid Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization to telemedicine follow-up versus routine in-person follow-up for the 1 week assessment after low-risk oculoplastic surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Patients in the telemedicine arm will have their post-operative week one visit via a telemedicine portal.
  Interventions: Other: Telemedicine follow-up
- Routine (No Intervention): Patient in the routine arm will have their post-operative week one visit in clinic.

INTERVENTIONS:
Other: Telemedicine follow-up — A telemedicine follow-up form based in REDCap that collects information from the patient including: history, photographs, vision measurement, and questions.
  Arms: Telemedicine

SUMMARY:
The investigators propose utilizing a simple telemedical protocol to allow patients to substitute the first post-operative visit with a remote survey that includes essential post-operative history, vision measurement, and photographs, all of which can be provided using a personal computer, tablet, or smart phone. The investigators have selected for this purpose a subset of oculoplastic procedures involving the eyelid and lacrimal system that have well-reported low rates of serious complications, since high-risk procedures will likely always require close, in-person care. The investigators hypothesize that telemedicine follow-up for the first post-operative week after low-risk oculoplastic surgery will decrease the time burden on patients without compromising their satisfaction or increase the risk of late post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Are age 18 years or older
* Are fluent in English
* Own or have ready access to a smart phone, tablet, or personal computer with high speed internet
* Participate in an informed consent process with the surgeon(s) including documentation of written informed consent
* Are undergoing a low-risk* eyelid procedure in a clinic, ambulatory surgery center, or hospital operating room setting, including but not limited to:

  * upper eyelid blepharoplasty repair
  * ectropion repair
  * entropion repair
  * external levator resection
  * internal levator resection
  * eyelid lesion removal and/or biopsy
  * eyelid reconstruction and defect repair including after Mohs' surgery
  * eyelid tightening procedures for Floppy Eyelid Syndrome
  * tarsorrhaphy
  * dacryocystorhinostomy

(*)These listed procedures have a low reported rate of serious complications including vision loss, infection, severe bleeding, or death; however, surgical risk is ultimately determined by the surgeon on a per-patient basis, except in those cases specifically excluded in the subsequent section.

Exclusion Criteria:

* Are under the age of 18 years
* Are incarcerated
* Are pregnant or plan to become pregnant during the period of surgery and 3 month recovery (however these patients are not eligible for elective eyelid surgery)
* Are not fluent in English
* Do not have access to or do not feel comfortable using a smart phone, tablet, or personal computer
* Lack personal capacity for consent (i.e. those patients requiring consent for the surgery by a legal representative are excluded)
* Experience a serious intra-operative complication (this criterion is assessed after initial consent)
* Are undergoing eyelid or other oculoplastic procedures that are deemed greater than low-risk for serious complications, including but not limited to:

  * orbital surgery
  * lower eyelid blepharoplasty
  * repair of extensive eyelid defects following Mohs' surgery (roughly >33%)
  * procedures requiring skin grafting
  * procedures requiring extensive tissue rearrangement
  * procedures involving an implant (e.g. frontalis sling, gold weight implantation; except dacryocystorhinostomy due to the low-risk nature of the lacrimal stent)
  * procedures requiring in-person care at the first post-operative week (e.g. suture removal, bolster removal, patch removal)

Notably, patients undergoing greater than low risk procedures listed here are absolutely excluded from this trial. Surgeon assessment of individual patient surgical risk only applies to those typically low-risk procedures listed in the previous section on inclusion criteria; reasons for escalation of risk level include patient characteristics (e.g. frailty, previous infection or wound dehiscence), re-operation/revision status, or other factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
FACE-Q 'Satisfaction with Outcome' | Approximately 3 months post-operatively
  A patient-reported outcome measure assessing satisfaction with the surgical outcome.

SECONDARY OUTCOMES:
FACE-Q 'Early Life Impact' | Approximately 1 week post-operatively
  A patient-reported outcome measure assessing early life impact of facial plastic surgery.
FACE-Q 'Satisfaction with Doctor' | Approximately 3 months post-operatively
  A patient-reported outcome measure assessing satisfaction with the surgeon.
Late post-operative complications | Between the first and second post-operative visits (approximately 1 week to 3 months)
  Investigator-reported post-operative complications.
Time burden | Approximately 1 week post-operatively
  Patient-reported time spent on the first post-operative visit, including waiting, travel, the visit, and all forms.

CONTACTS AND LOCATIONS:
Overall Officials: Davin C Ashraf, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Only plan to share in the event that journal requests de-identified data to be released.

REFERENCES:
- [Background] Vyas KS, Hambrick HR, Shakir A, Morrison SD, Tran DC, Pearson K, Vasconez HC, Mardini S, Gosman AA, Dobke M, Granick MS. A Systematic Review of the Use of Telemedicine in Plastic and Reconstructive Surgery and Dermatology. Ann Plast Surg. 2017 Jun;78(6):736-768. doi: 10.1097/SAP.0000000000001044. PMID 28328635
- [Background] Hwa K, Wren SM. Telehealth follow-up in lieu of postoperative clinic visit for ambulatory surgery: results of a pilot program. JAMA Surg. 2013 Sep;148(9):823-7. doi: 10.1001/jamasurg.2013.2672. PMID 23842982
- [Background] Kummerow Broman K, Roumie CL, Stewart MK, Castellanos JA, Tarpley JL, Dittus RS, Pierce RA. Implementation of a Telephone Postoperative Clinic in an Integrated Health System. J Am Coll Surg. 2016 Oct;223(4):644-51. doi: 10.1016/j.jamcollsurg.2016.07.010. Epub 2016 Aug 18. PMID 27545100
- [Background] Robaldo A, Rousas N, Pane B, Spinella G, Palombo D. Telemedicine in vascular surgery: clinical experience in a single centre. J Telemed Telecare. 2010;16(7):374-7. doi: 10.1258/jtt.2010.091011. Epub 2010 Aug 2. PMID 20679407
- [Background] Williams AM, Bhatti UF, Alam HB, Nikolian VC. The role of telemedicine in postoperative care. Mhealth. 2018 May 2;4:11. doi: 10.21037/mhealth.2018.04.03. eCollection 2018. PMID 29963556
- [Background] Carter SR, Stewart JM, Khan J, Archer KF, Holds JB, Seiff SR, Dailey RA. Infection after blepharoplasty with and without carbon dioxide laser resurfacing. Ophthalmology. 2003 Jul;110(7):1430-2. doi: 10.1016/S0161-6420(03)00447-0. PMID 12867404
- [Background] Chang S, Lehrman C, Itani K, Rohrich RJ. A systematic review of comparison of upper eyelid involutional ptosis repair techniques: efficacy and complication rates. Plast Reconstr Surg. 2012 Jan;129(1):149-157. doi: 10.1097/PRS.0b013e318230a1c7. PMID 22186506
- [Background] Lee EW, Holtebeck AC, Harrison AR. Infection rates in outpatient eyelid surgery. Ophthalmic Plast Reconstr Surg. 2009 Mar-Apr;25(2):109-10. doi: 10.1097/IOP.0b013e3181994124. PMID 19300151
- [Background] Mejia JD, Egro FM, Nahai F. Visual loss after blepharoplasty: incidence, management, and preventive measures. Aesthet Surg J. 2011 Jan;31(1):21-9. doi: 10.1177/1090820X10391212. PMID 21239669
- [Background] Kam KY, Cole CJ, Bunce C, Watson MP, Kamal D, Olver JM. The lateral tarsal strip in ectropion surgery: is it effective when performed in isolation? Eye (Lond). 2012 Jun;26(6):827-32. doi: 10.1038/eye.2012.34. Epub 2012 Mar 9. PMID 22402697